CLINICAL TRIAL: NCT04119544
Title: Intensive Rehabilitation Program With Intensive Visual Numerical Simulation Device for Improving Distal Motor Performance and Upper Limb Functional Capacity in Subacute Hemiparetics After Stroke. Randomized Controlled Trial.
Brief Title: Mirror Therapy Rehabilitation of the Upper Limb After Stroke (NEURO-MIROIR 2)
Acronym: NEUROMIROIR2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Les Trois Soleils (Other)
Collaborators: Clinalliance Villiers-sur-Orge (Unknown); Centre de Rééducation Fonctionnelle Pasori (Unknown); CHU de Reims (Other); Clinique Les Grands Chênes (Unknown); Clinique Napoléon (Unknown); Clinique Mariénia (Unknown); Clinique Verdaich (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-A00966-51
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: stroke; mirror therapy; rehabilitation; hemiparesis; upper limb; function; motor control
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Rehabilitation (Active Comparator): at least 4 sessions/week for 6 weeks, from 1 hour of conventional upper limb rehabilitation by an occupational therapist.
  Interventions: Other: Conventional rehabilitation
- Intensive Visual Simulation (Experimental): at least 4 sessions/week for 6 weeks, of 1 hour of upper limb rehabilitation including 45 minutes of conventional rehabilitation (occupational therapy) and 15 minutes of work with a medical device allowing intensive visual digital simulation.
  Interventions: Other: Conventional rehabilitation; Device: Intensive Visual Simulation

INTERVENTIONS:
Other: Conventional rehabilitation — upper limb rehabilitation involving submaximal passive amplitude stretching movements, inhibition postures, active efforts assisted of varying difficulty, target approach exercises with or without elbow support and gripping tasks, adapted to the upper limb's paresis abilities. The patient will be encouraged to gradually dispense with the assistance provided by the therapist or any technical assistance (suspension...) and thus to carry out the exercises in free active as soon as possible.
Device: Intensive Visual Simulation — * First week: observation, mentalization and then attempt to perform the movements on the screen.
  * Second and third weeks: production of analytical movements of wrist flexion/extension, pronation/supination, finger flexion/extension, thumb opposition.
  * From the 4th week until the end: depending on the patient's motor capacities, continuation of the work of the previous 2 weeks or introduction of more functional work with object manipulation, gripping work.
  Conventional rehabilitation upper limb rehabilitation involving submaximal passive amplitude stretching movements, inhibition postures, active efforts assisted of varying difficulty, target approach exercises with or without elbow support and gripping tasks, adapted to the upper limb's paresis abilities. The patient will be encouraged to gradually dispense with the assistance provided by the therapist or any technical assistance (suspension...) and thus to carry out the exercises in free active as soon as possible.
  Arms: Intensive Visual Simulation

SUMMARY:
Hemiparesis is a common motor disorder after a stroke. The majority of patients do not recover functional use of their paretic upper limb.

The use of mirror therapy allows the activation of the mirror neurons involved to stimulate brain plasticity after brain damage.The IVS (Intensive Visual Stimulation) device allows an easy implementation of mirror therapy by filming the valid upper limb and projecting the inverted image onto a screen placed above the parietal arm thus producing the illusion of movement of the parietal arm.

The main hypothesis of this study is that the structured practice of a large number of upper limb targeted movement repetitions using an intensive visual numerical simulation device as a partial replacement for routine care (conventional occupational therapy) in the sub-acute phase of stroke will increase the active function (motor function and functional abilities) of the distal end of the upper limb compared to conventional rehabilitation.

Objectives: This randomized controlled trial will evaluate the effects of partial substitution of routine care (occupational therapy) by structured movement repetition programs by Intensive Visual Simulation using an IVS3 device, on the distal motor control of the upper hemiparesis limb, between 4 and 10 weeks after the stroke, compared to a program with conventional care alone.

DETAILED DESCRIPTION:
Hemiparesis is a common motor disorder after a stroke. The majority of patients do not reuse their paretic upper limb.

Hypothesis: The structured practice of repeating upper limb movements by Intensive Visual Simulation will increase distal motor control, and improve the objective functional abilities of the upper limb.

Main Objective:Evaluate in a controlled protocol the effects, on the distal motor control of the upper hemiparesis limb, between 4 and 10 weeks after stroke, of 6 weeks of partial substitution of routine care (occupational therapy) by structured movement repetition programs by Intensive Visual Simulation using an IVS3 device, compared to 6 weeks of a program involving only conventional rehabilitation care, in a population of moderate to severe hemiparesis stroke patients in subacute phase.

Device Description: The IVS3 (Intensive Visual Simulation) rehabilitation device, marketed by Dessintey, allows the implementation of intensive mirror therapy by making it more immersive, ergonomic, and accessible. The IVS3 device consists of a hollow table adjustable in height, a touch screen dedicated to the therapist to set up the device and a large screen adjustable in height and sliding laterally to overlap the upper limb and thus allow the illusion that the limb visible on the screen is the paretic upper limb.

Methods: Multicentric randomised controlled Trial.

Risk/Constraint: To our knowledge, this research does not involve any risks other than those of daily life. The medical device will be used under normal conditions of use as described in the user manual. No contraindications are specified for this device. A risk of discomfort may be felt by the patient during the first few minutes of use. Possibility of feeling tired.

Research duration : 8 years Duration of patient participation : 18 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Stroke hemiparesis on unilateral focal lesion dating from 4 to 10 weeks at baseline;
* Total sub-scores wrist and hand of th Fugl-Meyer < 16
* Patient having agreed to sign an informed consent
* patient being affiliated to the French Social Security

Exclusion Criteria:

* Cognitive dysfunction or progressive intercurrent illness making effective communication or participation in the study impossible
* Phasic disorders that prevent the understanding of instructions
* Patient include in an other clinical trial
* Neurological conditions prior to stroke
* Patient who had mirror therapy or IVS rehabilitation before inclusion
* Rheumatological pathology of the hand and wrist
* Person under legal protection measure.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of motor performance score on the Fugl-Meyer sub-score wrist/hand | between Day1(day of program start), Week6 (end of the program)
  Fugl-Meyer (FM) assessment for measures of the motor impairment of the upper-limb; the sub-score wrist/hand includes items related to movements of the forearm (proximal arm), wrist, hand (distal arm) and speed/coordination during a finger-nose task. The total sub-score range between 0 and 30.

SECONDARY OUTCOMES:
Change of motor performance score on the Fugl-Meyer | between Day1(day of program start), Week6 (end of the program) and Week18 (12 weeks after the end of the program)
  Fugl-Meyer (FM) assessment for measures of the motor impairment of the upper-limb; the test includes items related to movements of the shoulder, elbow, forearm (proximal arm), and wrist and hand (distal arm). The total scores range between 0 and 66.
Change of motor capacity on Stroke Upper Limb Capacity Scale (SULCS) | between Day1(day of program start), Week6 (end of the program) and Week18 (12 weeks after the end of the program)
  The scale measures active upper limb capacity in hemiparesis based on 10 items, with each item having a possible score of 0 or 1. Three items for arm capacity without active hand capacity, four items for arm capacity and basic hand capacity and three items for complex hand capacity.The total scores range between 0 and 10.
Change of spasticity score of the elbow flexors, wrist flexors, finger flexors measured by the Modified Ashworth Scale (MAS) | between Day1(day of program start), Week6 (end of the program) and Week18 (12 weeks after the end of the program)
  The Modified Ashworth scale (MAS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. Scoring :0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the Range Of Movement (ROM)
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Change in perceived stroke impact on the Stroke Impact Scale (SIS) | between Day1(day of program start), Week6 (end of the program) and Week18 (12 weeks after the end of the program)
  The Stroke Impact Scale (SIS) is a 59 item patient reported outcome measure, covering 8 domains: strength (4 items), hand function (5 items), mobility (9 items), activities of daily living (10 items), memory (7 items), communication (7 items), emotion (9 items), and handicap (8 items). Domains are scored on a metric of 0 to 100, with higher scores indicating better self-reported health. Four of the scales of the SIS can be combined into a composite physical domain (strength, hand function, physical and instrumental activities of daily living, and mobility), with scores also presented on a 0 to 100 metric.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe DURET, MD, Principal Investigator — Clinique Les Trois Soleils; Manuel Wiese, MD, Principal Investigator — Clinalliance Villiers-sur-Orge; Nikolay DOBREV, MD, Principal Investigator — CRF PASORI; François BOYER, Professor, Principal Investigator — Hôpital Sébastopol, CHU de Reims; Caroline TERRACOL, MD, Principal Investigator — Clinique Marienia Inicea; Jean-Marc GUEBLE, MD, Principal Investigator — Clinique Verdaich; Adrien PETIT, MD, Principal Investigator — Clinique Les Grands Chênes Inicea; Magali CAPLANNE, MD, Principal Investigator — Clinique Napoléon Inicea
Locations (5):
- France (5):
  - CHU Sébastopol, Reims, Champagne-Ardenne
  - Clinique Napoléon, Saint-Paul-lès-Dax, Nouvelle-Aquitaine
  - Clinique Les Trois Soleils, Boissise-le-Roi
  - CRF Pasori, Cosne-Cours-sur-Loire
  - Clinalliance Villiers-sur Orge, Villiers-sur-Orge